CLINICAL TRIAL: NCT01872273
Title: Blood Cell Response to Exercise
Status: Withdrawn | Type: Observational
Why Stopped: Project never funded. No subjects were recruited.
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC026
Record Dates: First submitted 2013-05-01; First posted 2013-06-07 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Obese; Overweight; Hypertension; Hyperlipidemia; Glucose Intolerant; High blood sugar; Exercise in obesity; Platelets
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Overweight; Hypertension; Hyperlipidemias; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Moderate Physical Exercise — This intervention is comprised of two separate visits at least one week apart. The purpose of visit 1 is to determine the cycle ergometer workload that produces a moderate exercise intensity of 60% heart rate reserve to be used on visit 2. The purpose of visit 2 is to determine changes in platelet reactivity in response to moderate exercise.

SUMMARY:
Moderate exercise is recommended to improve cardiovascular health in obese and overweight people particularly with metabolic syndrome (MetS) that have hypertension, elevated fasting blood sugar, and elevated blood lipids. This study is being done to determine how platelets respond when a person performs an initial period of moderate exercise.

ELIGIBILITY:
Inclusion Criteria:

* 30-60 years old
* BMI >/=26 and <40 kg/m2
* not planning to or currently attempting to gain or lose weight
* low reported omega-3 fatty acid intake per Omega-3 Checklist
* Metabolic Syndrome as define 3/5 of the following:Waist circumference: men > 102 cm women > 88 cm, triglycerides > 150 mg/dL, HDL cholesterol: men < 40 mg/dL women < 50 mg/dL,Blood pressure >130/>85 mmHg,Fasting glucose > 100 mg/dL (Hypertensive subjects are eligible if taking thiazide diuretics NOT ACE inhibitors beta blockers)

Exclusion Criteria:

* smoke or use tobacco or nicotine in any form (including pills and patches)
* take any medication that makes you unable to exercise
* have established cardiovascular, pulmonary, and/or metabolic disease such as diabetes
* have uncontrolled hypertension
* have alcohol, anabolic steroid, or other substance abuse issues
* consume more than 3 alcoholic drinks/week
* have joint or muscle injuries that affects your ability to exercise
* have cancer (other than skin cancer or carcinoma in situ of the cervix
* pregnant or lactating
* currently exercise regularly
* taking non-steroidal anti-inflammatory medications (aspirin, Aleve, Advil, ibuprofen, naproxen
* take lipid modifying medications such as statins (Lipitor, Zocor)
* take medications for blood glucose such as insulin or metformin
* take medications that affect platelet functions (Plavix)
* taking omega-3 supplements (fish or flax oil)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese adults with Metabolic Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity | Baseline, post-intervention (24 hours), & time points during the exercise phase: prior to exercise (-25 min, -10 min, - 1 min), 10 minutes into the routine, at completion (25 minutes), and 20 & 60 minutes following completion
  We hypothesize that moderate physical exercise will increase platelet reactivity in sedentary individuals with metabolic syndrome. Platelet reactivity will be measured by flow cytometry using anti-CD61 antibodies as a marker for platelets and anti-CD62 (P-selectin) as a marker of platelet activation. This will be measured at baseline, post-intervention and time points post-baseline in each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center

IPD SHARING:
Plan to Share IPD: No